CLINICAL TRIAL: NCT02051348
Title: A Single-blinded, Placebo Controlled, Crossover Study of Pylopass Versus Placebo in Subjects Who Are Helicobacter Pylori Carriers and With Mild Indigestion
Brief Title: Study of Pylopass Versus Placebo in Subjects Who Are Helicobacter Pylori Carriers and With Mild Indigestion
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Atlantia Food Clinical Trials (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AFCRO-046
Record Dates: First submitted 2014-01-30; First posted 2014-01-31 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: HELICOBACTER INFECTION
Keywords: Helicobacter pylori; Mild Indigestion
MeSH Terms: conditions — Helicobacter Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo - 2 doses per day for 4 weeks
  Interventions: Biological: Pylopass; Biological: Placebo
- Pylopass (Active Comparator): Probiotic - 2 doses per day for 4 weeks
  Interventions: Biological: Pylopass; Biological: Placebo

INTERVENTIONS:
Biological: Pylopass — Pylopass
Biological: Placebo — Placebo

SUMMARY:
Helicobator pylori (H. pylori) is a bacteria which survives in the lining of the stomach. An estimated 50% of the world's population is infected with H. pylori. Developing economies, such as in Southeast Asia, the Indian subcontinent and Latin America, have prevalence rates of as high as 90%.

H. pylori infection often goes undiagnosed, as many sufferers do not experience any adverse symptoms. Infection with H. pylori is described as "not a disease in itself but a condition that affects the relative risk of developing various clinical disorders of the upper gastrointestinal tract.' Clinically relevant symptoms could include peptic ulcer, melena or secondary conditions such as iron deficiency anemia or vitamin B12 deficiency.

There is evidence that probiotics can be beneficial for those with gastrointestinal diseases. Pylopass contains the probiotic strain Lactobacillus reuteri, which was selected for its anti-H. pylori characteristics and in clinical trials has shown to result in a reduction in urease breath test values in subjects with H. pylori.

The objective of this study is to evaluate the ability of Pylopass to reduce H. pylori load in subjects who are H. pylori positive.

DETAILED DESCRIPTION:
Helicobator pylori (H. pylori) is a gram negative, spiral shaped bacteria which colonizes in the gastric mucosa. An estimated 50 percent of the world's population is infected with H. pylori.

H. pylori infection does not necessarily result in clinically relevant symptoms. Ching and Wong report that most cases of H. pylori are asymptomatic . Moreover, Kusters et al states that infection with H. pylori "is not a disease in itself but a condition that affects the relative risk of developing various clinical disorders of the upper gastrointestinal tract" (Kusters, 2006). Clinically relevant symptoms could include peptic ulcer, melena or secondary conditions such as iron deficiency anemia or vitamin B12 deficiency.

The most recent iteration of the Maastricht/Florence Consensus report outlines the diagnostic guidelines and treatment strategies for those with H. pylori (Malfertheiner 2012). Individuals with certain risk factors, such as a family history of gastric cancer, bleeding ulcer or with secondary disease such as iron deficiency anemia should undergo eradication therapy. For those with functional dyspepsia, the test and treat strategy has been recommended. However, there remains a lack of options for volunteers who are either asymptomatic or experience mild gastrointestinal symptoms who are not indicated for eradication therapy or to undergo the test and treat strategy.

There is evidence that probiotics can be beneficial for those with gastrointestinal diseases. A review by Ritchie and Romanuk succinctly summarizes this point by writing that "probiotics are generally beneficial in treatment and prevention of gastrointestinal diseases" (Ritchie 2012). In the context of H. pylori infection, probiotics are administered alongside conventional eradication treatment regimens to lessen the severity of side effects and improve tolerance. Francavilla et al has studied the impact of Lactobacillus reuteri on H. pylori load levels, as measured by urea breath test (UBT) values. The researchers found that a significant reduction in H. pylori load as evidenced by significantly decreased UBT values. They also found a decrease in symptom scores as measured by the Gastrointestinal Symptom Rating Scale (GSRS) (Francavilla 2008). Imase et al has also studied the impact of Lactobacillus reuteri supplementation in H. pylori infected individuals and found a suppressive effect from the L. reuteri tablets on UBT values (Imase 2007). These studies indicate that Lactobacillus reuteri exerts an effect on H. pylori by lowering the load.

There are many potential mechanisms by which probiotic strains, such as Lactobacillus reuteri, could exert a suppressive effect against H. pylori. One potential method is to stabilize or strengthen the gut mucosal barrier. Other mechanisms include sequestration of H. pylori, production of antimicrobial substances or through competitive binding to receptors in the gut (Garcia, 2009; Lesbros-Pantoflickova, 2007).

The Pylopass strain of Lactobacillus reuteri (L. reuteri) was identified after a detailed, multi-year screening process. It was selected for its anti-H. pylori characteristics from a culture collection of 8,000 different food grade strains. The original commensal environment of the Pylopass strain of L. reuteri is from humans. L. reuteri is considered one of the few autochthonous lactobacilli in humans and animals known to the scientific community. It has been isolated in the gastrointestinal tract of humans, pigs, cattle and dogs (Casas 2000). It has also been isolated in a variety of different foods, such as milk products and fermented rice noodles.

Pylopass is comprised of Lactobacillus reuteri cells, suspended in a matrix and spray dried. As such, the Lactobacillus reuteri cells are metabolically inactive. However, through in vitro and human studies, it has been shown to exert an H. pylori load lowering effect. In vitro work has found that Pylopass specifically coaggregates with H. pylori under acidic conditions. Two human pilot studies have shown that oral administration of Pylopass leads to a reduction in UBT values in volunteers with H. pylori (Mehling 2013). As the cells of the Lactobacillus reuteri in Pylopass do not need to be metabolically active to exert a benefical effect, this provides tremendous advantages in developing economies, where there are many cases of antibiotic resistant H. pylori.

The advantages of Pylopass over other Lactobacillus products are product stability, specificity for H. pylori and stability in gastric conditions. As previously mentioned, the highest prevalence of H. pylori is in developing economies, where access to an adequate cold chain may not be reliable. As Pylopass is comprised of inactivated cells which can withstand environmental fluctuations, it is appropriate for shipments that do not require temperature control. Secondly, while probiotics cater to general gut health, Pylopass specifically bind H. pylori under acidic conditions. Thirdly, the mechanism of action is not dependent on binding sites or survival in the gastric environment. Probiotics can be beneficial because they may replace harmful bacteria in the gastrointestinal tract. However, it is uncertain whether such living strains can withstand the acidic environment in the stomach. This concern is not a challenge for Pylopass as the coaggregation depends only on the binding of surface structures between Pylopass and H. pylori. As there are advantages to Pylopass over traditional probiotic strains, it is the goal of this study to confirm that the results from the first two human trials hold true.

Given the challenges of rising rates of antibiotic resistance, delivery of a product which is relevant and useful in developing economies, development of a product which can withstand environmental fluctuations and the lack of options for H. pylori positive individuals who are not indicated for eradication therapy, the development of Pylopass could be an important tool to address these challenges. To this end, the goal of this study is to assess the impact of a four week supplementation period of Pylopass on markers of Helicobacter pylori load in volunteers who do not meet the full criteria for eradication therapy as outlined by the Maastricht Florence Consensus report.

The primary outcome of this study is the urease breath test (UBT), a widely validated non-invasive measure for H. pylori status. However, we also recognize that there are limitations of using the urease breath test. The primary limitation is that the UBT serves as a proxy measure for Helicobacter pylori load levels and does not provide direct assessments of the health of the gastric mucosa or of H. pylori load. By including a subset of volunteers for gastric biopsies, the degree of inflammation can be directly assessed and the H pylori load can be quantified. By performing biopsies at two time points, before and after supplementation with the active ingredient, the effects of the supplement on the health of the gastric mucosa can be assessed. Due to the small subset of volunteers, the information will be qualitative in nature, but will provide a scientific basis for assessing participants in future studies. As antibiotic resistance is on the rise in cases of Helicobacter pylori, it is important to continuously develop new adjunctive solutions which may help improve the health of the gastric mucosa, and the best way to assess this directly is through the use of gastric biopsies.

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible for enrolment into the study, subjects must;

1. Be able to give written informed consent,
2. Be between 18 and 75 years of age,
3. Be in generally good health as determined by the investigator OR have mild gastrointestinal discomfort, such as mild indigestion,
4. Have a positive urease breath test (> 1.5)

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the below criteria;

1. Are less than 18 and greater than 75 years of age,
2. Females are pregnant, lactating or wish to become pregnant during the study.
3. Are hypersensitive to any of the components of the test product,
4. Have a significant acute or chronic, unstable and untreated disease or any condition which contraindicates, in the investigators judgement, entry to the study,
5. Have an active gastrointestinal disorder or previous gastrointestinal surgery,
6. Having a condition or have taken a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results; to include proton pump inhibitors or gastroprotective medicines,
7. Have taking antibiotics in the past 3 months,
8. Prior eradication therapy with antibiotics for H. pylori infection,
9. Have not made any major dietary changes in the past 3 months,
10. Are taking non-steroidal anti-inflammatory drugs (NSAIDs) within 2 weeks of baseline visit or for the duration of the trial,
11. History of illicit drug use,
12. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial,
13. Subjects may not be receiving treatment involving experimental drugs,
14. If the subject has been in a recent experimental trial, these must have been completed not less than 60 days prior to this study,
15. Have a malignant disease or any concomitant end-stage organ disease,

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of Pylopass to reduce H pylori load by urease breath test (UBT) | Up to 8 weeks

SECONDARY OUTCOMES:
Symptoms, using the Gastrointestinal Symptom Rating Scale (GSRS) | Up to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martin JM Buckley, MRCPI, FRCPI, Principal Investigator — Mercy University Hospital
Locations (1):
- Atlantia Food Clinical Trials, University College Cork, Cork, Ireland

REFERENCES:
- [Derived] Buckley M, Lacey S, Doolan A, Goodbody E, Seamans K. The effect of Lactobacillus reuteri supplementation in Helicobacter pylori infection: a placebo-controlled, single-blind study. BMC Nutr. 2018 Dec 7;4:48. doi: 10.1186/s40795-018-0257-4. eCollection 2018. PMID 32153909